CLINICAL TRIAL: NCT06978816
Title: Auricular Acupoint Embedding as Adjunctive Therapy to NSAIDs for Accelerated Relief of Renal Colic in Urolithiasis: A Randomized Controlled Trial
Brief Title: Ear Pressure Points Plus Pain Meds for Faster Kidney Stone Pain Relief
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gao Xiaofeng (Other)
Responsible Party: Sponsor-Investigator, Gao Xiaofeng, Senior Attending Urologist, Changhai Hospital, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHC2025-130
Record Dates: First submitted 2025-04-27; First posted 2025-05-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-05

CONDITIONS: Renal Colic; Acupuncture, Ear
Keywords: Kidney Calculi; Renal Colic; acupuncture, ear
MeSH Terms: conditions — Renal Colic; Kidney Calculi | interventions — Anti-Inflammatory Agents, Non-Steroidal; Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum Auricular Acupoint Embedding Group (Experimental): In the experimental group, patients received verum auricular acupoint embedding using disposable sterile press needles (0.22×0.5 mm) at three ipsilateral ear points - thalamus (MA-AT), kidney (MA-SC), and shenmen (MA-TF1) - combined with intravenous infusion of 50 mg dexketoprofen trometamol (a non-steroidal anti-inflammatory drug) as adjuvant therapy.
  Interventions: Drug: Non-Steroidal anti-inflammatory drugs (NSAIDS); Other: Auricular Acupoint Embedding
- Sham Auricular Acupoint Embedding Group (Sham Comparator): In the control group, participants received sham auricular stimulation using non-penetrating adhesive patches applied to the same ipsilateral ear points (thalamus [MA-AT], kidney [MA-SC], and shenmen [MA-TF1]) without needle insertion, combined with identical intravenous administration of 50 mg dexketoprofen trometamol (NSAID) as per the experimental protocol
  Interventions: Drug: Non-Steroidal anti-inflammatory drugs (NSAIDS); Other: Sham Acupoint Embedding

INTERVENTIONS:
Drug: Non-Steroidal anti-inflammatory drugs (NSAIDS) — Intravenous infusion of 50 mg dexketoprofen trometamol injection
Other: Auricular Acupoint Embedding — Concurrently with the intravenous infusion of dexketoprofen trometamol, verum auricular acupoint embedding was performed using disposable sterile press needles at three ipsilateral ear points: thalamus (MA-AT), kidney (MA-SC), and shenmen (MA-TF1), with needle retention for 60 minutes
  Other Names: acupuncture, ear
  Arms: Verum Auricular Acupoint Embedding Group
Other: Sham Acupoint Embedding — Concurrently with the intravenous infusion of dexketoprofen trometamol, sham auricular stimulation was administered using non-penetrating adhesive patches applied to three ipsilateral ear points: thalamus (MA-AT), kidney (MA-SC), and shenmen (MA-TF1), maintaining the application for 60 minutes.
  Arms: Sham Auricular Acupoint Embedding Group

SUMMARY:
Title: Can Ear Acupressure Help Relieve Kidney Stone Pain Faster When Combined with Painkillers?

Purpose:

This study tests whether adding ear acupressure to standard painkillers (NSAIDs) helps adults with kidney stone pain feel better faster. The investigators also want to know if this combination causes any side effects.

Key Questions:

Does ear acupressure + NSAIDs reduce pain more quickly than NSAIDs alone? Are there any safety concerns with this treatment? How does real ear acupressure compare to a fake (placebo) procedure? Who Can Join? Adults aged 18-75 Experiencing moderate-to-severe kidney stone pain (confirmed by CT or ultrasound) No recent painkiller use or allergies to NSAIDs

What Participants Will Do:

Receive in the emergency room:

Real treatment: Tiny needles placed on 3 ear points + NSAIDs (ketorolac injection) OR Placebo treatment: Fake tape on ear points + NSAIDs (same injection) Rate their pain on a 0-10 scale over 60 minutes. Have their heart rate and blood pressure checked.

Study Details:

Duration: Single ER visit (no long-term follow-up) Participants Needed: 116 Safety: Rescue pain medication (like morphine) is available if needed.

Why This Matters:

Kidney stones cause severe pain, and current painkillers may not work fast enough. Ear acupressure is a low-risk method from traditional Chinese medicine that could provide quicker relief.

Ethics:

Approved by Changhai Hospital's Ethics Committee. Participants can leave the study anytime.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15 and 75 years (inclusive)
2. Diagnosis of urinary tract stones confirmed by CT or ultrasound
3. Visual Analog Scale (VAS) score ≥ 4 (indicating moderate to severe renal colic)
4. No severe cardiac, hepatic, or pulmonary dysfunction, and no coagulation disorders.
5. No psychiatric disorders

Exclusion Criteria:

1. Use of any analgesic medication within the past 6 hours.
2. Allergy to NSAIDs, morphine, or anisodamine (scopolamine derivatives)
3. History of asthma, urticaria, congestive heart failure, acute ischemic heart disease, acute cerebrovascular disease, or increased intracranial pressure
4. Active peptic ulcer, pyloric obstruction, or intestinal obstruction
5. Severe adverse reactions to acupuncture in the past
6. Pregnancy or lactation
7. Unwillingness to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Response rate of Visual Analog Scale (VAS) reduction | At 0, 5, 10, 15, 20, 30, 45, and 60 minutes after intervention initiation
  The Visual Analog Scale (VAS) is a validated, subjective measurement tool widely used in clinical research to assess symptom intensity (e.g., pain, nausea). It consists of a 100-mm horizontal or vertical line anchored by two extremes: "no symptom" (0 mm) and "worst imaginable symptom" (100 mm). Participants mark their current level of intensity, with the score determined by measuring the distance from the "no symptom" endpoint.Response rate of Visual Analog Scale (VAS) reduction (defined as ≥50% decrease from baseline)

SECONDARY OUTCOMES:
Recurrence rate of pain within 48 hours | Within 48 hours after the completion of this emergency treatment
  "Recurrence" is defined as revisiting the emergency department due to renal colic.
Incidence of adverse reactions | At 0, 5, 10, 15, 20, 30, 45, and 60 minutes after intervention initiation
  Adverse reactions refer to harmful effects caused by medical treatment, such as: nausea, rash, dizziness, abnormal liver function, etc.
body temperature | At 0, 5, 10, 15, 20, 30, 45, and 60 minutes after intervention initiation
  Body temperature refers to the internal temperature of the human body and is a key indicator for maintaining normal physiological functions and metabolic activities. It is typically measured in degrees Celsius (°C) or Fahrenheit (°F), and its stable range is precisely regulated by the hypothalamus (the body's thermoregulatory center).
Blood pressure | At 0, 5, 10, 15, 20, 30, 45, and 60 minutes after intervention initiation
  Blood pressure refers to the force exerted by circulating blood against the walls of blood vessels, primarily the arteries. It is conventionally measured in mmHg. It is a vital physiological parameter that ensures adequate blood flow to organs and tissues.
Heart rate | At 0, 5, 10, 15, 20, 30, 45, and 60 minutes after intervention initiation
  Heart rate refers to the number of heartbeats per minute (bpm), reflecting the cardiac cycle frequency. It is a vital cardiovascular parameter indicating circulatory system function.

IPD SHARING:
Plan to Share IPD: Undecided